Table of Planned Analyses
Breathe with Ease: A Unique Approach to Managing Stress (BEAMS)
PI: Stephen J. Teach, MD, MPH
Final 11.25.16

| Symptom-free days In last 14 days; symptom-free days are defined as a 24-hour period with no coughing, wheezing, chest tightness, or shortness of breath and no need for rescue medications Secondary Outcomes Asthma morbidity In last 14d: daytime/nighttime symptoms, activity limitation, use of quick relief meds, changed plans, and missed school. Asthma medication adherence Medication use in past 2d Medication use lin past 2d Medication use lin past 2d Medication use prevents exacerbations) ED visits, hospital admissions, ICU admissions, ICU admissions, ICU admissions, Primary care visits Asthma exacerbations Perceived Stress Scale Stressful Life Events Parental stress Perceived Stress Scale Stressful Life Events Parental depression CES-D Child anxiety PROMIS Parent Proxy Depressive Symptoms Quality of life Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) Safety data Asis/SAEs Exploratory Outcomes Coping strategies Brief COPE Mindfulness Interpersonal mindfulness of parenting Parental Resilience Control Variables Baseline Sociodemographic factors Age, gender, race, ethnicity, insurance type, parent education, household income, family medical history, parent health literacy, parental resilience factors Intervention uptake, satisfaction, and fidelity Asthma severity NAEPP classification, as determined by IMPACT DC clinician | Primary Outcome | |
|---|---|---|
| Asthma morbidity Asthma medication Asthma medication Asthma medication Asthma medication Adherence Medication use in past 2d Medication beliefs (difficulty following med plan, concerns re side effects belief that med use prevents exacerbations) Health care utilization Feature in the properties of the properties o | Symptom-free days | <ul> <li>In last 14 days; symptom-free days are defined as a 24-hour period with<br/>no coughing, wheezing, chest tightness, or shortness of breath and no<br/>need for rescue medications</li> </ul> |
| relief meds, changed plans, and missed school. Asthma medication adherence • Medication use in past 2d • Medication beliefs (difficulty following med plan, concerns re side effects belief that med use prevents exacerbations) • ED visits, • hospital admissions, • ICU admissions, • primary care visits Asthma • exacerbations Asthma • Courses of systemic steroids or hospitalizations in 12m prior to enrollment and during 12m follow up period (independent courses ≥7d apart) Parental stress • Perceived Stress Scale • Stressful Life Events Parental depression • PROMIS Parent Proxy Anxiety Child anxiety • PROMIS Parent Proxy Depressive Symptoms Quality of life • Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) Safety data • AEs/SAEs Exploratory Outcomes Coping strategies • Brief COPE Mindfulness • Interpersonal mindfulness of parenting Parental Resilience • LOT-R Economic data • Analysis of costs of care in both groups Environmental smoke exposure • Parent smoking behavior Use of existing ancillary services • Participation in stress reducing activities (exercise, dance, yoga, breathing, other) Control Variables Baseline Sociodemographic factors Intervention uptake, satisfaction, and idelity Asthma severity • NAEPP classification, as determined by IMPACT DC clinician | | |
| adherence • Medication beliefs (difficulty following med plan, concerns re side effects belief that med use prevents exacerbations) • ED visits, • hospital admissions, • ICU admissions, • primary care visits Asthma exacerbations • Courses of systemic steroids or hospitalizations in 12m prior to enrollment and during 12m follow up period (independent courses ≥7d apart) Parental stress • Perceived Stress Scale • Stressful Life Events Parental depression Child anxiety • PROMIS Parent Proxy Anxiety Child depression Child depression Child anxiety • PROMIS Parent Proxy Depressive Symptoms Quality of life • Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) Safety data • AEs/SAEs Exploratory Outcomes Coping strategies Mindfulness • Interpersonal mindfulness of parenting Parental Resilience Economic data • Analysis of costs of care in both groups • Child smoke exposure Parental mode exposure • Parent smoking behavior Use of existing ancillary services • Participation in stress reducing activities (exercise, dance, yoga, breathing, other) Control Variables Baseline Sociodemographic factors Intervention uptake, satisfaction, and fidelity Asthma severity • NAEPP classification, as determined by IMPACT DC clinician | , | |
| <ul> <li>hospital admissions,</li> <li>ICU admissions,</li> <li>primary care visits</li> <li>Courses of systemic steroids or hospitalizations in 12m prior to enrollment and during 12m follow up period (independent courses ≥7d apart)</li> <li>Parental stress</li> <li>Perceived Stress Scale</li> <li>Stressful Life Events</li> <li>Parental depression</li> <li>CES-D</li> <li>Child anxiety</li> <li>PROMIS Parent Proxy Anxiety</li> <li>Child depression</li> <li>PROMIS Parent Proxy Depressive Symptoms</li> <li>Quality of life</li> <li>Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ)</li> <li>Safety data</li> <li>AEs/SAEs</li> <li>Exploratory Outcomes</li> <li>Coping strategies</li> <li>Brief COPE</li> <li>Mindfulness</li> <li>Interpersonal mindfulness of parenting</li> <li>Parental Resilience</li> <li>LOT-R</li> <li>Economic data</li> <li>Analysis of costs of care in both groups</li> <li>Environmental smoke exposure</li> <li>Parent smoking behavior</li> <li>Use of existing ancillary services</li> <li>Use of mental health resources</li> <li>Participation in stress reducing activities (exercise, dance, yoga, breathing, other)</li> <li>Control Variables</li> <li>Baseline Sociodemographic factors</li> <li>Intervention uptake, satisfaction, and fidelity</li> <li>Age, gender, race, ethnicity, insurance type, parent education, household income, family medical history, parent health literacy, parental resilience sessions, use of stress management techniques, use of techniques with children</li> <li>NAEPP classification, as determined by IMPACT DC clinician</li> </ul> | adherence | Medication beliefs (difficulty following med plan, concerns re side effects, |
| exacerbations enrollment and during 12m follow up period (independent courses ≥7d apart) Parental stress • Perceived Stress Scale • Stressful Life Events Parental depression CES-D Child anxiety • PROMIS Parent Proxy Anxiety Child depression Quality of life • Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) Safety data • AEs/SAEs Exploratory Outcomes Coping strategies • Brief COPE Mindfulness Parental Resilience • LOT-R Economic data • Analysis of costs of care in both groups Environmental smoke exposure smoke exposure • Parent smoking behavior Use of existing ancillary services • Participation in stress reducing activities (exercise, dance, yoga, breathing, other) Control Variables Baseline Sociodemographic factors Intervention uptake, satisfaction, and fidelity Asthma severity • NAEPP classification, as determined by IMPACT DC clinician | Health care utilization | <ul><li>hospital admissions,</li><li>ICU admissions,</li></ul> |
| Stressful Life Events Parental depression CES-D Child anxiety PROMIS Parent Proxy Anxiety Child depression Quality of life Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) Safety data AEs/SAEs Exploratory Outcomes Coping strategies Mindfulness Parental Resilience Economic data Environmental smoke exposure Use of existing ancillary services Baseline Sociodemographic factors Intervention uptake, satisfaction, and fidelity Asthma severity Stressful Life Events CES-D PROMIS Parent Proxy Anxiety Proxy Anxiety PROMIS Parent Proxy Anxiety PROMIS Parent Proxy Anxiety PROMIS Parent Proxy Anxiety PROMIS Parent Proxy Anxiety Proxy Anxiety PACQLQ AEs/SAEs Exploratory Outcomes Coping strategies Parent Sches Parent Sches Parent Smoking behavior Parent smoking behavior Use of existing ancillary services Parent smoking behavior Use of psychological support (parent/child/other family members) Use of mental health resources Parent smoking behavior Use of psychological support (parent/child/other family members) Use of mental health resources Parent smoking behavior Use of psychological support (parent/child/other family members) Use of mental health resources Parent smoking behavior Use of psychological support (parent/child/other family members) Use of psychological support (parent/child/other family members) Control Variables Baseline Sociodemographic factors Intervention uptake, satisfaction, and fidelity Age, gender, race, ethnicity, insurance type, parent education, household income, family medical history, parent health literacy, parental resilience | | enrollment and during 12m follow up period (independent courses ≥7d |
| Child anxiety Child depression Quality of life Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) Safety data AEs/SAEs Exploratory Outcomes Coping strategies Mindfulness Parental Resilience Economic data Environmental smoke exposure Use of existing ancillary services Baseline Sociodemographic factors Baseline Sociodemographic factors Intervention uptake, satisfaction, and fidelity Asthma severity PROMIS Parent Proxy Anxiety PROMIS Parent Proxy Depressive Symptoms PROMIS Parent Proxy Depressive Symptoms PROMIS Parent Proxy Depressive Symptoms PROMIS Parent Proxy Depressive Symptoms Proxy Depressive Symptoms Pacuality of Life Questionnaire (PACQLQ) Intervention youtcomes Corping strategies Brief COPE Intervention uptake, satisfaction, and fidelity Asthma severity Pacintary Proxy Depressive Symptoms Pacuality Proxy Depressive Symptoms Pacuality Proxy Depressive Symptoms Pacuality Proxy Depressive Symptoms Pacuality of Life Questionnaire (PACQLQ) Pacuality of Life Questionnaire (Pacuality of Life Questionnaire (Pacuality of Life Questionnaire (Pacuality of Life Questionnaire (Pacua | Parental stress | |
| Child depression Quality of life Safety data Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) Safety data AEs/SAEs Exploratory Outcomes Coping strategies Mindfulness Parental Resilience Economic data Environmental smoke exposure Use of existing ancillary services Baseline Baseline Baseline Baseline Control Variables Baseline Intervention uptake, satisfaction, and fidelity Asthma severity Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) AEs/SAEs Exploratory Outcomes Brief COPE Interpersonal mindfulness of parenting AEs/SAEs Brief COPE Interpersonal mindfulness of parenting Corte LOT-R Child smoke exposure Parent smoking behavior Use of psychological support (parent/child/other family members) Use of mental health resources Participation in stress reducing activities (exercise, dance, yoga, breathing, other) Control Variables Age, gender, race, ethnicity, insurance type, parent education, household income, family medical history, parent health literacy, parental resilience Completion of 1:1 session, completion of group sessions, location/format of sessions, use of stress management techniques, use of techniques with children NAEPP classification, as determined by IMPACT DC clinician | Parental depression | CES-D |
| Child depression Quality of life Quality of life Safety data AEs/SAEs Exploratory Outcomes Coping strategies Mindfulness Parental Resilience Economic data Environmental smoke exposure Use of existing ancillary services Baseline Sociodemographic factors Intervention uptake, satisfaction, and fidelity Asthma severity Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) AEs/SAEs Brief COPE Intervention yutcomes Intervention uptake, satisfaction, and fidelity NAEPP classification, as determined by IMPACT DC clinician | Child anxiety | PROMIS Parent Proxy Anxiety |
| Safety data Exploratory Outcomes Coping strategies Mindfulness Parental Resilience Economic data Environmental smoke exposure Use of existing ancillary services Baseline Sociodemographic factors Intervention uptake, satisfaction, and fidelity Asthma severity Parent Smoke Spinal Parent Smoking Spinal Spina | Child depression | |
| Exploratory Outcomes | Quality of life | Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) |
| Coping strategies Mindfulness Parental Resilience Economic data Environmental smoke exposure Use of existing ancillary services Baseline Sociodemographic factors Intervention uptake, satisfaction, and fidelity Asthma severity • Brief COPE • Interpersonal mindfulness of parenting • LOT-R • LOT-R • Analysis of costs of care in both groups • Child smoke exposure • Parent smoking behavior • Use of psychological support (parent/child/other family members) • Use of mental health resources • Participation in stress reducing activities (exercise, dance, yoga, breathing, other) Control Variables Age, gender, race, ethnicity, insurance type, parent education, household income, family medical history, parent health literacy, parental resilience Completion of 1:1 session, completion of group sessions, location/format of sessions, use of stress management techniques, use of techniques with children • NAEPP classification, as determined by IMPACT DC clinician | Safety data | AEs/SAEs |
| <ul> <li>Mindfulness</li> <li>Interpersonal mindfulness of parenting</li> <li>Parental Resilience</li> <li>LOT-R</li> <li>Economic data</li> <li>Analysis of costs of care in both groups</li> <li>Environmental smoke exposure</li> <li>Child smoke exposure</li> <li>Parent smoking behavior</li> <li>Use of existing ancillary services</li> <li>Use of mental health resources</li> <li>Participation in stress reducing activities (exercise, dance, yoga, breathing, other)</li> <li>Control Variables</li> <li>Baseline Sociodemographic factors</li> <li>Intervention uptake, satisfaction, and fidelity</li> <li>Asthma severity</li> <li>NAEPP classification, as determined by IMPACT DC clinician</li> </ul> | | |
| Parental Resilience Economic data • Analysis of costs of care in both groups Environmental smoke exposure • Child smoke exposure • Parent smoking behavior Use of existing ancillary services • Participation in stress reducing activities (exercise, dance, yoga, breathing, other) Control Variables Baseline Sociodemographic factors Intervention uptake, satisfaction, and fidelity Asthma severity • LOT-R • Analysis of costs of care in both groups • Child smoke exposure • Parent smoking behavior • Use of psychological support (parent/child/other family members) • Use of mental health resources • Participation in stress reducing activities (exercise, dance, yoga, breathing, other) Control Variables Age, gender, race, ethnicity, insurance type, parent education, household income, family medical history, parent health literacy, parental resilience Completion of 1:1 session, completion of group sessions, location/format of sessions, use of stress management techniques, use of techniques with children Asthma severity • NAEPP classification, as determined by IMPACT DC clinician | Coping strategies | Brief COPE |
| Economic data • Analysis of costs of care in both groups • Child smoke exposure • Parent smoking behavior Use of existing ancillary services • Use of psychological support (parent/child/other family members) • Use of mental health resources • Participation in stress reducing activities (exercise, dance, yoga, breathing, other) Control Variables Baseline Sociodemographic factors Intervention uptake, satisfaction, and fidelity Asthma severity • Analysis of costs of care in both groups • Child smoke exposure • Parent smoking behavior • Use of psychological support (parent/child/other family members) • Use of mental health resources • Participation in stress reducing activities (exercise, dance, yoga, breathing, other) • Control Variables Control Variables Age, gender, race, ethnicity, insurance type, parent education, household income, family medical history, parent health literacy, parental resilience Completion of 1:1 session, completion of group sessions, location/format of sessions, use of stress management techniques, use of techniques with children • NAEPP classification, as determined by IMPACT DC clinician | Mindfulness | Interpersonal mindfulness of parenting |
| <ul> <li>Environmental smoke exposure</li> <li>Darent smoking behavior</li> <li>Use of existing ancillary services</li> <li>Use of psychological support (parent/child/other family members)</li> <li>Use of mental health resources</li> <li>Participation in stress reducing activities (exercise, dance, yoga, breathing, other)</li> <li>Control Variables</li> <li>Baseline Sociodemographic factors</li> <li>Intervention uptake, satisfaction, and fidelity</li> <li>Asthma severity</li> <li>Child smoke exposure</li> <li>Parent smoking behavior</li> <li>Use of psychological support (parent/child/other family members)</li> <li>Use of psychological support (parent/child/other family members)</li> <li>Use of psychological support (parent/child/other family members)</li> <li>Parent smoking behavior</li> <li>Use of psychological support (parent/child/other family members)</li> <li>Use of psychological support (parent/child/other family medical support (parent/child/other family members)</li> <li>Use of psychological support (parent/child/other family medical support (parent/child/other family members)</li> <li>Use of psychological support (parent/child/other family members)</li> <li>Use of psychological support (parent/child/other family members)</li> <li>Use of psychological support (parent/child/other family members)</li> &lt;</ul> | Parental Resilience | LOT-R |
| <ul> <li>Smoke exposure</li> <li>Use of existing ancillary services</li> <li>Use of psychological support (parent/child/other family members)</li> <li>Use of mental health resources</li> <li>Participation in stress reducing activities (exercise, dance, yoga, breathing, other)</li> <li>Control Variables</li> <li>Baseline Sociodemographic factors</li> <li>Intervention uptake, satisfaction, and fidelity</li> <li>Asthma severity</li> <li>Parent smoking behavior</li> <li>Use of psychological support (parent/child/other family members)</li> <li>Use of mental health resources</li> <li>Participation in stress reducing activities (exercise, dance, yoga, breathing, page page page page page page page page</li></ul> | Economic data | Analysis of costs of care in both groups |
| Use of existing ancillary services • Use of psychological support (parent/child/other family members) • Use of mental health resources • Participation in stress reducing activities (exercise, dance, yoga, breathing, other) Control Variables Baseline Sociodemographic factors Intervention uptake, satisfaction, and fidelity Asthma severity • Use of psychological support (parent/child/other family members) • Use of mental health resources • Participation in stress reducing activities (exercise, dance, yoga, breathing, other) Control Variables Age, gender, race, ethnicity, insurance type, parent education, household income, family medical history, parent health literacy, parental resilience sessions, use of stress management techniques, use of techniques with children Asthma severity • NAEPP classification, as determined by IMPACT DC clinician | | |
| <ul> <li>Use of mental health resources</li> <li>Participation in stress reducing activities (exercise, dance, yoga, breathing, other)</li> <li>Control Variables</li> <li>Baseline Sociodemographic factors</li> <li>Intervention uptake, satisfaction, and fidelity</li> <li>Asthma severity</li> <li>Use of mental health resources</li> <li>Participation in stress reducing activities (exercise, dance, yoga, breathing, other)</li> <li>Age, gender, race, ethnicity, insurance type, parent education, household income, family medical history, parent health literacy, parental resilience factors</li> <li>Completion of 1:1 session, completion of group sessions, location/format of sessions, use of stress management techniques, use of techniques with children</li> <li>NAEPP classification, as determined by IMPACT DC clinician</li> </ul> | - | • |
| Baseline Sociodemographic factors Intervention uptake, satisfaction, and fidelity Asthma severity Age, gender, race, ethnicity, insurance type, parent education, household income, family medical history, parent health literacy, parental resilience factors Completion of 1:1 session, completion of group sessions, location/format of sessions, use of stress management techniques, use of techniques with children NAEPP classification, as determined by IMPACT DC clinician | | <ul> <li>Use of mental health resources</li> <li>Participation in stress reducing activities (exercise, dance, yoga,</li> </ul> |
| Baseline Sociodemographic factors Intervention uptake, satisfaction, and fidelity Age, gender, race, ethnicity, insurance type, parent education, household income, family medical history, parent health literacy, parental resilience Completion of 1:1 session, completion of group sessions, location/format of sessions, use of stress management techniques, use of techniques with children Asthma severity Age, gender, race, ethnicity, insurance type, parent education, household income, family medical history, parent health literacy, parental resilience sessions, location/format of sessions, use of stress management techniques, use of techniques with children Asthma severity NAEPP classification, as determined by IMPACT DC clinician | 0 | |
| Sociodemographic factors Intervention uptake, satisfaction, and fidelity Asthma severity income, family medical history, parent health literacy, parental resilience factors, parental resilience income, family medical history, parent health literacy, parental resilience factors Completion of 1:1 session, completion of group sessions, location/format of sessions, use of stress management techniques, use of techniques with children NAEPP classification, as determined by IMPACT DC clinician | | |
| satisfaction, and fidelity sessions, use of stress management techniques, use of techniques with children Asthma severity • NAEPP classification, as determined by IMPACT DC clinician | Sociodemographic factors | income, family medical history, parent health literacy, parental resilience |
| | satisfaction, and | sessions, use of stress management techniques, use of techniques with |
| | | NAEPP classification, as determined by IMPACT DC clinician |
| NAEPP classification, as determined by impact DC clinician ACT score | Asthma control | NAEPP classification, as determined by IMPACT DC clinician |

Table of Planned Analyses
Breathe with Ease: A Unique Approach to Managing Stress (BEAMS)
Pl: Stephen J. Teach, MD, MPH

Final 11.25.16

We will examine interactions between primary and secondary outcomes and

- baseline asthma variables (severity/control, health care utilization, exacerbations),
- baseline psychosocial variables (parental stress and depression, resilience, child anxiety and depression, quality of life)
- baseline demographic factors

In addition, we will examine interactions between primary and secondary outcomes and intervention uptake within the intervention group.

Key planned analyses include:

- Interaction between primary outcome and parental age, education, household income, child age and gender
- Interaction between primary outcome and baseline child asthma severity, control, and history of unscheduled healthcare utilization
- Interaction between primary outcome and baseline parental depression
- Interaction between primary outcome and baseline parental stress
- Interaction between primary outcome and baseline parental resilience
- Interaction between primary outcome and baseline child depression
- Interaction between primary outcome and baseline child anxiety
- Interaction between primary outcome and baseline asthma severity/control
- Dose-response analysis of intervention uptake (session completion and parent report of technique utilization)

Sample Size Calculation: The sample size was recalculated on September 14, 2015 based on the baseline data collected from the first 60 participants, which showed the following:

- mean = 10.25 days
- standard deviation = 4.12
- median = 11.5 days.

The sample distribution is not normal and approximated a Poisson distribution. Based on this distribution, the calculated sample size is 188 to achieve 80% power at a 0.05 significance level to detect a response rate ratio of 1.15 with baseline response rate of 10.25. Therefore, with 10% percent attrition rate, we planned to enroll 207 participants.

The primary analyses for this study will be conducted at 6m FU, and the same analyses will be completed with the 12m FU data.

The primary analysis for this study will be by intention to treat.

A per-protocol analysis will also be conducted. Per protocol will be defined as completion of all four one-on-one sessions.